CLINICAL TRIAL: NCT01141296
Title: Randomized Controlled Study of Fenofibrate in Combination With Ursodeoxycholic Acid in Primary Biliary Cirrhosis
Brief Title: Fenofibrate in Combination With Ursodeoxycholic Acid (UDCA) in Primary Biliary Cirrhosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Miami (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cynthia Levy, MD, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Feno-01
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fenofibrate (Active Comparator)
  Interventions: Drug: fenofibrate
- sugar pill (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fenofibrate — fenofibrate 200 mg PO daily for 1 year
  Arms: Fenofibrate
Drug: placebo — Placebo pill identical to active drug will be given PO once a day for 1 year
  Arms: sugar pill

SUMMARY:
The purpose of this study is to determine if the combination of ursodeoxycholic acid (UDCA) and fenofibrate is more effective than UDCA alone in the treatment of primary biliary cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 and ≤ 75 years old
2. Established diagnosis of PBC and positive AMA
3. Previous treatment with UDCA 13-15 mg/kg/day for at least 1 year
4. Incomplete response to UDCA defined as serum ALP ≥ 2 times the upper limit of normal on two separate measurements despite at least 1 year of therapy with UDCA
5. Female patients of childbearing age need a negative pregnancy test performed within 7 days of enrollment, and need to be on adequate contraception throughout the study period
6. Signed informed consent after careful review of information and study details

Exclusion Criteria:

1. Hypersensitivity to fenofibrate
2. Administration of the following drugs at any time during the 3 months prior to screening for the study: methotrexate, colchicines, azathioprine, systemic steroids.
3. Prisoners and institutionalized subjects, pregnant or nursing women
4. Anticipated need for liver transplantation within one year (estimated 1-year survival <80% as predicted by the Mayo risk score).
5. Recipients of liver transplantation
6. Recurrent variceal hemorrhage, uncontrolled encephalopathy or refractory ascites
7. Co-existing liver diseases such as acute or chronic viral hepatitis, alcoholic liver disease, choledocholithiasis, autoimmune hepatitis, biopsy-proven non-alcoholic fatty liver disease, Wilson's disease and hemochromatosis
8. Acute or chronic renal failure, defined as GFR < 60 ml/min
9. Known history of cholecystitis with intact gallbladder
10. History of, or known high risk for, venous thromboembolism
11. Current use of warfarin or statins

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04

PRIMARY OUTCOMES:
Serum alkaline phosphatase level | one year

SECONDARY OUTCOMES:
Symptoms - quality of life | one year
  Quality of life will be evaluated throught the NIDDK questionnaire at entry and end of study
symptoms - pruritus | one year
  Pruritus will be evaluated through a visual analogue scale and the 5-D questionnaire, both applied at entry and end of study
symptom -fatigue | one year
  fatigue will be evaluated through the Fatigue Impact Scale applied at entry and end of study
interleukin 1 | one year
  IL-1 will be measured from stored serum collected at entry and end of study. This will be measured by Beadlyte Human Multicytokine Detection system.
interleukin 6 | one year
  IL-6 will be measured from stored serum collected at entry and end of study. This will be measured by Beadlyte Human Multicytokine Detection system.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Levy, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota